CLINICAL TRIAL: NCT02208791
Title: Evaluation of the Effects of Sirolimus Addition to the Triple Immunosuppression Protocol on Peripheral Blood Lymphocytes and Development of Anti-HLA Antibodies in Sensitized Kidney Transplant Recipients - a Pilot Study
Brief Title: Effects of the Quadruple Immunosuppression on Peripheral Blood Lymphocytes and Development of Anti-HLA Antibodies in Kidney Transplant
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U1111-1157-7462
Record Dates: First submitted 2014-08-01; First posted 2014-08-05 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2014-06

CONDITIONS: Kidney Transplantation
Keywords: Kidney Transplantation; Graft Rejection; Immunossupression
MeSH Terms: interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tacrolimus/MPS/Prednisone (Active Comparator): This arm will be maintained with current conventional triple immunosuppression. Sirolimus will not be added to this arm
  Interventions: Drug: No intervention
- Sirolimus/Low Tacrolimus/MPS/Prednisone (Experimental): Sirolimus, 2mg once daily, will be added to the maintenance immunosuppression composed of tacrolimus, prednisone and mycophenolate. The prescription of tacrolimus will be tapered down to achieve a peripheral blood trough level between 3 e 5 ng/mL and micophenolate will be reduced to 540mg bid..
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — Sirolimus, 2mg once daily, will be added to the maintenance immunosuppression composed of tacrolimus, prednisone and mycophenolate. The prescription of tacrolimus will be tapered down to achieve a peripheral blood trough level between 3 e 5 ng/mL and micophenolate will be reduced to 540mg bid.
  Arms: Sirolimus/Low Tacrolimus/MPS/Prednisone
Drug: No intervention
  Arms: Tacrolimus/MPS/Prednisone

SUMMARY:
The purpose of this study is to determine the effects of sirolimus in the phenotype of peripheral blood T and B lymphocytes regarding their naïve, memory, effector end regulatory phenotype and in the development of anti-HLA antibodies among kidney transplant recipients with high immunological risk for graft rejection.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, ages 18 to 60 years inclusive
* Percentage of Panel Reactive Antibodies at transplantation > 20%
* Estimated glomerular filtration rate using MDRD formula at inclusion >29ml/min

Exclusion Criteria:

* Subjects with a history of cancer
* Subjects with a previous non kidney transplantation
* Subjects receiving any immunosuppression different of tacrolimus/prednisone/mycophenolate
* Subjects with a urinary protein/creatinine ratio greater than 0.3
* Subjects with active HBV, HCV and HIV infection

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2014-07; Primary Completion 2016-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
A composite of graft loss and/or death with graft function | up to one year

SECONDARY OUTCOMES:
Number of participants with serious and non-serious adverse events and the incidence of biopsy proven acute allograft rejection | Up to one year

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital das Clinicas - Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo, Brazil